CLINICAL TRIAL: NCT05619211
Title: Improving Cardiorespiratory Fitness and Cardiometabolic Health Among Children With Physical Disabilities Through Movement-to-Music Telehealth With Arm-based Sprint-Intensity Interval Training
Brief Title: Piloting Movement-to-Music With Arm-based Sprint-Intensity Interval Training Among Children With Physical Disabilities
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Byron Lai, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300010372; 1R21HD109358-01A1 (NIH)
Record Dates: First submitted 2022-11-02; First posted 2022-11-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Movement-to-Music (Experimental): 12 weeks of sprint-intensity interval training while following along with YouTube videos that include arm-based routines, with coaching through telecommunications. Participants are instructed to maintain their habitual diet and nutrition patterns
  Interventions: Behavioral: Sprint-Intensity Interval Training with Telecoaching
- Wait-list Control (No Intervention): 12 weeks of maintaining habitual physical activity, diet, and nutrition patterns, until receiving 12 weeks of Movement-to-Music

INTERVENTIONS:
Behavioral: Sprint-Intensity Interval Training with Telecoaching — Maximal intensity exercises that use the arms.
  Arms: Movement-to-Music

SUMMARY:
This study is investigating the potential effects of a high-intensity home-exercise program among children with cerebral palsy. The program includes rhythmic movements to music that are adapted for wheelchair uses and age-appropriate themes. This project has the potential to address a large knowledge gap in the extant literature, because there are no widely accessible, evidence-based, enjoyable, and age-appropriate modalities for improving cardiovascular fitness or cardiometabolic health among children with disabilities who have mobility disabilities.

ELIGIBILITY:
We are recruiting 50 parent-child dyads. Childs are the participant undergoing the exercise intervention. Parents are required to support the safety and schedule of the child participant. Parents are considered participants due to their responsibilities.

Inclusion Criteria:

* have a medical diagnosis of cerebral palsy, as determined by ICD-10 codes
* aged 6-17 years old
* a Gross Motor Function Classification System Level I-IV (as determined via participant screening, explained in the protocol section below)
* medical clearance to participate in high-intensity exercise from a physician (using the attached medical screening form and explained in the intervention safety, monitoring, and response plan)
* access to a Wi-Fi Internet connection in the home via mobile phone or tablet computer
* a caregiver who will support and monitor the participant's safety during the intervention and manage the child's exercise schedule.

Exclusion Criteria:

* physically active (defined as >150 minutes per week of self-reported moderate-to-vigorous intensity exercise in a typical week)
* cannot use their arms for exercise
* a Gross Motor Function Classification Level of V
* complete blindness or deafness;
* Any past history of a contraindication to exercise testing according to American College of Sports Medicine (ACSM) guidelines (Liguori and American College of Sports Medicine, 2020): significant change in the resting electrocardiogram suggesting significant ischemia, myocardial infarction, or other cardiac event, unstable angina, uncontrolled cardiac dysrhythmias causing symptoms or hemodynamic compromise, symptomatic severe aortic stenosis, uncontrolled symptomatic heart failure, pulmonary embolus or pulmonary infarction, myocarditis or pericarditis, aneurysm.
* pregnant (due to radiation from a Dual Energy X-ray Absorptiometry [DEXA] scan)
* has not been seen by a physician within the last year
* uses a g-tube

Eligible caregivers will include parents or legal guardians of the child, who can commit sufficient time to support the child in their roles for the study and communicate in English. Caregivers who have complete blindness or deafness will be excluded from participation.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2023-09-29 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Changes in pVO2 | Week 0, Week 13
  peak oxygen consumption (mL/kg-1/min-1) obtained from a graded exercise test on an arm ergometer

SECONDARY OUTCOMES:
change in body weight | Week 0, Week 13
  body weight in pounds (lbs) measured via DXA scan
changes in total body fat | Week 0, Week 13
  body fat in pounds (lbs) measured via DXA scan
changes in total lean mass | Week 0, Week 13
  lean mass in pounds (lbs) measured via DXA scan
changes in lean tissue percentage | Week 0, Week 13
  percentage of lean tissue per whole body weight
changes in fat tissue percentage | Week 0, Week 13
  percentage of fat tissue per whole body weight
changes in C-reactive protein | Week 0, Week 13
  hsCRP (mg/L) measured via dried blood spot test
changes in Hemoglobin A1C | Week 0, Week 13
  HbA1C (mmol/mol) measured via dried blood spot test
changes in fasting insulin | Week 0, Week 13
  Fasting Insulin (μIU/mL) measured via dried blood spot test
changes in fasting triglycerides | Week 0, Week 13
  Fasting Triglycerides (mg/dL) measured via dried blood spot test
changes in fasting high-density lipoprotein | Week 0, Week 13
  HDL cholesterol (mg/dL) measured via dried blood spot test
changes in fasting low-density lipoprotein | Week 0, Week 13
  LDL cholesterol (mg/dL) measured via dried blood spot test
Changes in systolic blood pressure | Week 0, Week 13
  systolic blood pressure (mmHg) measured via blood pressure cuff
Changes in diastolic blood pressure | Week 0, Week 13
  diastolic blood pressure (mmHg) measured via blood pressure cuff

OTHER OUTCOMES:
Adherence to the exercise prescription | Week 1 - 12
  Percentage of video minutes completed versus prescribed
Perceived Enjoyment | Week 0, Week 13
  Physical Activity Enjoyment Scale (PACES). The scale ranges from 0 to 48. Scores above 24 are considered high enjoyment while being physically active.
Recruitment, enrollment, and attrition rates | Week 1 - 12
  Percentage of those who do the above, divided by the total participants
Adverse events | Week 1 - 12
  Any adverse event reported by participants

CONTACTS AND LOCATIONS:
Locations (1):
- Wellness Health And Research Facility (WHARF), Homewood, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be submitted into the NICHD Data and Specimen Hub (DASH). Intellectual property and data generated under this project will be administered in accordance with both University and NIH policies, including the NIH Data Sharing Policy and Implementation Guidance under notice NOT-OD-03-032 (released February 26, 2003)
Supporting Information: Study Protocol
Time Frame: Beginning 3 months after publication and ending 5 years after publication.

REFERENCES:
- [Derived] Lai B, Oster RA, Davis D, Bright L, Fisher G, Wilroy J, Kim Y, Young R, Wright A, Sinha T, Rimmer JH. Telehealth Movement-to-Music With Arm-Based Sprint-Intensity Interval Training to Improve Cardiometabolic Health and Cardiorespiratory Fitness in Children With Cerebral Palsy: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2024 Mar 5;13:e56499. doi: 10.2196/56499. PMID 38441939